CLINICAL TRIAL: NCT04385563
Title: A Phase III,Randomized,Multicenter,Double-blind Clinical Trail to Evaluate the Efficacy,Safety and Immunogenicity of the Combination of TQ-B211 Plus Docetaxel Versus Herceptin® Plus Docetaxel as First-line Treatment in Patients With HER2-positive MBC.
Brief Title: A Study to Evaluate the Efficacy and Safety of the Combination of TQ-B211 Plus Docetaxel in Patients With HER2-positive MBC.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TQB211-III-01
Record Dates: First submitted 2020-05-09; First posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: HER2-positive Metastatic Breast Cancer
MeSH Terms: interventions — Trastuzumab; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TQ-B211 + docetaxel (Experimental): Participants will be administered TQ-B211 plus docetaxel once every three weeks(Q3W) in cycles up to cycle 8.
  Interventions: Drug: TQ-B211; Drug: docetaxel
- Herceptin®+docetaxel (Active Comparator): Participants will be administered Herceptin® plus docetaxel Q3W in cycles up to cycle 8.
  Interventions: Drug: Herceptin®; Drug: docetaxel

INTERVENTIONS:
Drug: TQ-B211 — Participants will receive TQ-B211 8 milligrams/kilogram (mg/kg) intravenously(iv.) on day 1 in Cycle 1 followed by 6 mg/kg iv.on day 1 in Cycles 2 to 8.
  Arms: TQ-B211 + docetaxel
Drug: Herceptin® — Participants will receive Herceptin® 8 milligrams/kilogram (mg/kg) intravenously(iv.) on day 1 in Cycle 1 followed by 6 mg/kg iv.on day 1 in Cycles 2 to 8.
  Arms: Herceptin®+docetaxel
Drug: docetaxel — Participants will receive docetaxel 75 milligrams/square meter (mg/m^2) iv.on day 2 in Cycle 1 followed by 75mg/m^2 iv.on day 1 in Cycles 2 to 8.

SUMMARY:
To evaluate the efficacy,safety and immunogenicity of TQ-B211 plus docetaxel versus Herceptin® plus docetaxel in Patients with HER2-positive metastatic breast cancer.Trastuzumab plus docetaxel was chosen as the comparator in the control group,as it represents a common first-line treatment option used in HER2+ MBC population in China.

ELIGIBILITY:
Inclusion Criteria:

* Ability to give written informed consent.
* Age：≥18 and ≤75,female.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1；Life expectancy of at least 12 weeks.
* Histologically confirmed diagnosis as her2-positive metastatic or locally recurrent breast cancer that cannot be treated with radical surgery or radiotherapy.
* No prior systematical chemotherapy, biotherapy or molecule-targeted therapy for metastatic breast cance.
* Patients must have a measurable disease according to RECIST v. 1.1 28 days before randomization. (Disease in brain or bone will not be included)
* Left ventricular ejection fraction (LVEF) ≥50 percent (%)
* Blood routine examination should meet the following conditions: Absolute neutrophil count (ANC)≥1.5×109/L Platelets ≥100 x 109/L Hemoglobin ≥90 g/L hemameba≥3.0×109/L )
* Liver function should meet the following conditions:

Total bilirubin ≤1.5x Upper Limit of Normal(ULN); Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤3x ULN if no liver involvement or ≤5x ULN with liver involvement.

-Kidney function should meet the following conditions: Cr (creatinine) ≤1.5x ULN or Ccr (creatinine clearance rate) ≥50 mL/min.

* The coagulation function should meet the following conditions: International normalized ratio（INR）≤1.5；Activated partial thromboplastin time or partial thromboplastin time ≤1.5×ULN
* Female who meet the following criteria can participate in the study:

No childbearing potential； Female with childbearing potential: negative pregnancy test within 7 days before the first administration of the investigational drug; patients are not breastfeeding; Contraception use must continue for the duration of study treatment and for at least 6 months after the last dose of study treatment.

Exclusion Criteria:

* Not eligible for docetaxel combination therapy.
* Endocrine therapy within 2 weeks before randomization.
* Patients had received neoadjuvant or adjuvant therapy with herceptin 12 months before randomization.
* Patients had received neoadjuvant/adjuvant drugs containing other anthracycline or taxol 6 months before randomization.
* Patients had used Chinese patent medicine or Chinese herbal medicine with anti-cancer activity 2 weeks before randomization.
* Brain metastases with symptom/untreated brain metastases/other central nervous system(CNS) metastases. Treated CNS metastases remain stable for at least 4 weeks before the study, and no evidence of cerebral edema, no sign for glucosinolates or anticonvulsants treatments.
* Patients with a previous malignancy within the past 5 years (other than curatively treated in situ carcinoma of the cervix, non-melanoma skin cancer and superficial bladder carcinoma).
* Hepatitis virus C(HCV) positive, HIV positive, syphilis positive, or HBsAg positive and Hepatitis virus B(HBV) DNA titer in peripheral blood is beyond the normal range.
* Patients had received major surgical procedures (including open chest biopsy) major trauma (e.g. fracture) within 4 weeks before randomization, and there are unhealed wounds, ulcers or fractures at the time of screening or major surgery is expected during the study
* Patients have a history of hypertensive encephalopathy or a hypertension or an uncontrolled hypertension ( systolic blood pressure >150mmHg or diastolic blood pressure >100mmHg with antihypertensive drugs)
* Patients had a history of myocardial infarction 6 months before randomization; medical history of congestive heart failure in New York heart association classification (NYHA)≥ grade II,and a severe arrhythmia that cannot be controlled by drugs（atrial fibrillation and paroxysmal supraventricular tachycardia are excluded）;LVEF had previously declined to less than 50% during or after new trastuzumab adjuvant or adjuvant therapy.
* Allergies to herceptin ®/ TQ-B211 or the chemotherapies involved in this trial and their excipients.
* History hypersensitivity to any study drug .
* Patients had participated in clinical trials of other antitumor drugs 4 weeks before randomization .
* Not eligible to join the study judged by investigators.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Estimated)
Dates: Start 2018-11-11 (Actual); Primary Completion 2021-02 (Estimated); Study Completion 2021-10 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Baseline up to week 24（Baseline up to 8 cycles）
  ORR was defined as percentage of participants with partial response (PR) or complete response (CR) determined on the basis of investigator assessments.

SECONDARY OUTCOMES:
Duration of Response (DOR) | up to week 120
  DOR was defined as the time from the date of initial confirmed PR or CR to the date of disease progression or death within the study.
Progression-free survival (PFS) | up to week 120
  PFS was defined as the time from randomization to the first occurrence of disease progression or death from any cause, whichever occurred first, on the basis of investigator assessments.
Disease control rate(DCR) | up to week 120
  DCR was defined as the percentage of participants with best overall response of CR, PR, stable disease (SD) and Non-CR/Non-progressive disease (PD).
Overall survival (OS) | up to week 120
  OS was defined as the time from the date of randomization to the date of death from any cause.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality